CLINICAL TRIAL: NCT01483521
Title: Externalizing Behavior in Early Childhood: A Randomized Control Evaluation of a Home Visitation Program
Brief Title: Infant Psychiatry Home Visitation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Childrens Hospital Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H08-02992
Record Dates: First submitted 2011-11-24; First posted 2011-12-01 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Aggression; Hyperactivity; Impulsive Behaviors
Keywords: Randomized; Home visitation; Externalizing disorder; Parenting stress; Childhood externalizing disorders; Positional defiant
MeSH Terms: conditions — Aggression; Spasm; Impulsive Behavior | interventions — House Calls; Psychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Waitlist families (Experimental): Experimental arm consisted of randomized waitlist families who received home visitation where mothers were taught to play with their children in a developmentally appropriate manner and also engaged in a co-construction task.
  Control arm families did not get any active intervention. Parents from both arm types completed pre and post questionnaires to measure child's externalizing behaviors and parenting stress.
  Parents from experimental group were encouraged to keep a diary of their play record.
  Interventions: Other: Clinical home visitation

INTERVENTIONS:
Other: Clinical home visitation — Clinical Home visitation consisted of once a month visits to families on the experimental group. During those visits home visitors facilitated developmentally appropriate play guidance and co-construction tasks for the dyad.
  Other Names: Home visiting; Externalizing disorders; Parenting stress

SUMMARY:
This is a proposed home visitation program for families of children with externalizing behaviors who are on the wait list for psychiatric assessment at BC Children's hospital. The aim of this program is to implement and evaluate a home visitation strategy in order to support those waiting up to four months to consult a psychiatrist.

DETAILED DESCRIPTION:
The Home visitation program was developed in response to long wait lists for the Infant Psychiatry Program. This home visitation program intervention consists of the following components: Developmental guidance, empowerment of parents while respecting the parent-child attachment, and child centered interactional guidance. The home visitors ( a PhD student and a Masters level student) visit consenting families and gave the parents an opportunity to voice their concerns regarding their child's behaviors. They were instructed to co-construct a play that had to be child led. Home visitors facilitated this task. Parents completed the Child Behavior Checklist and Parenting Stress Index prior to and after the intervention. These home visitations occurred approximately once a month whilst the families were on the wait list for clinical assessment and treatment. Those families that were randomized in control group did not receive any intervention.

Extended description of the protocol, including information not already contained in other fields.

ELIGIBILITY:
Inclusion Criteria:

* Children with externalizing disorders referred to Infant Psychiatry Clinic of Children's hospital and on the wait list

Exclusion Criteria:

* Children over 6 years old
* Children with internalizing disorder
* Families that reside outside of the Vancouver due to practicality of home visitation,
* Families requiring an interpreter

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Reduction of externalizing disorders and child's aggression | Participants will be followed for the duration of their time on the Clinic's wait list, an expected average of 10 weeks
  The specific units of measure to be assessed pre and post intervention are the mean scores of the CBCL (overall score, attention problems subscale, externalizing subscale, aggression subscale) and the PSI (overall score, parent distress sub scale, parent-child dysfunctional interaction, difficult child subscale).

SECONDARY OUTCOMES:
Measurement of parental stress | Participants will be followed for the duration of their time on the Clinic's wait list, an expected average of 10 weeks
  Measurement of parental stress after the intervention was offered

CONTACTS AND LOCATIONS:
Overall Officials: Pratibha Reebye, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada